CLINICAL TRIAL: NCT04987996
Title: Randomized Double-Blind Placebo Controlled Phase II Study of a Galectin Inhibitor (GR-MD-02) and Pembrolizumab Versus Pembrolizumab and Placebo in Patients With Metastatic Melanoma and Head and Neck Squamous Cell Carcinoma
Brief Title: GR-MD-02 + Pembrolizumab Versus Pembrolizumab Monotherapy in Melanoma and Squamous Cell Head and Neck Cancer Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn due to lack of supply of one of the investigational agents.
Sponsor: Providence Health & Services (Other)
Collaborators: Providence Cancer Center, Earle A. Chiles Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020000655
Record Dates: First submitted 2021-07-14; First posted 2021-08-03 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Melanoma; Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC; MM; pembrolizumab; GR-MD-02; Galectin Inhibitor; GRMD-02; GRMD002
MeSH Terms: conditions — Melanoma; Squamous Cell Carcinoma of Head and Neck | interventions — belapectin; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GR-MD-02 + pembrolizumab (Experimental): 4 mg/kg GR-MD-02 in combination with standard pembrolizumab treatment.
  Interventions: Drug: GR-MD-02; Drug: Pembrolizumab
- Pembrolizumab Monotherapy (Placebo Comparator): 4 mg/kg placebo in combination with standard pembrolizumab treatment.
  Interventions: Drug: Placebo; Drug: Pembrolizumab

INTERVENTIONS:
Drug: GR-MD-02 — Patients will receive up to seventeen doses of GR-MD-02 intravenously over 85 Days.
  Other Names: Galactoarabino-rhamnogalactouronate
  Arms: GR-MD-02 + pembrolizumab
Drug: Placebo — Patients will receive up to seventeen doses of placebo intravenously over 85 Days.
  Arms: Pembrolizumab Monotherapy
Drug: Pembrolizumab — Patients will receive 200mg doses of pembrolizumab intravenously over 85 Days.
  Other Names: Keytruda

SUMMARY:
The purpose of this study is to test the safety & efficacy of combination drugs versus placebo to treat metastatic melanoma and head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
Eligible patients will be registered, stratified by diagnosis (melanoma versus OHN cancer), and the number of prior systemic therapies, and randomized to receive either GR-MD-02 + pembrolizumab or pembrolizumab + placebo.

In addition to monitoring for toxicity and clinical response, blood and tumor samples will be obtained to assess immunologic measures relevant to galectin biology and pembrolizumab T-cell checkpoint inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable or metastatic melanoma including unknown primary, mucosal or uveal melanomas. Histological confirmation of melanoma will be required by previous biopsy or cytology. Patients with recurrent or metastatic head and neck squamous cell carcinoma (HNSCC) with disease progression during or after platinum-containing chemotherapy are eligible. PD-L1 testing is not needed for OHN cancers.
* Patients who have received anti-PD1 or anti-PD-L1 in the past are eligible if it has been at least 6 months since the last anti-PD-1 or PD-L1 dose, they meet all other eligibility criteria and progression of malignancy has been documented on imaging. Progression for this patient subset is defined as the appearance of one or more new metastatic sites, or a 5% or greater increase in the sum of diameter of target lesions or an unequivocal increase in non-target site. Treatment naïve melanoma patients are eligible.
* Patients must be ≥ 18 years of age.
* ECOG performance status of 0-2.
* Women of childbearing potential must have a serum or urine pregnancy test performed within 72 hours prior to the start of protocol treatment. The results of this test must be negative in order for the patient to be eligible. In addition, women of childbearing potential as well as male patients must agree to take appropriate precautions to avoid pregnancy.
* No active bleeding.
* Anticipated lifespan greater than 12 weeks.
* Patients must sign a study-specific consent document.

Exclusion Criteria:

* Patients who have previously received a galectin antagonist.
* Patients with active autoimmune disease except for autoimmune thyroiditis or vitiligo (see Appendix C).
* Patients with history of autoimmune colitis.
* Patients with untreated brain metastases. Patients with treated brain metastases who demonstrate control of brain metastases with follow-up imaging 4 or more weeks after initial therapy are eligible.
* Patients requiring other systemic oncologic therapy, including experimental therapies.
* Patients with active infection requiring antibiotics.
* Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus.
* Need for steroids at greater than physiologic replacement doses. Inhaled corticosteroids are acceptable.
* Laboratory exclusions (to be performed within 28 days of enrollment):

  * WBC < 3.0 x 109/L
  * Hgb < 9.0 g/dL
  * AST or ALT > 1.5 times ULN
  * Total bilirubin > 1.9 g/dL, unless due to Gilbert's Syndrome. If Gilbert's Syndrome is present by clinical history, then direct bilirubin must by < 3.0 g/dl.
  * Known history of HIV
  * Known history of Hepatitis B
  * Known history of Hepatitis C
  * INR > 1.5x ULN
* Inability to give informed consent and comply with the protocol. Patients must be judged able to understand fully the investigational nature of the study and the risks associated with the therapy.
* Any medical condition that in the opinion of the Principal Investigator would compromise the safety or conduct of the study procedures.
* Unresolved immune-mediated pneumonitis, diarrhea, elevation of hepatocellular enzymes or other toxicities requiring greater than physiological replacement doses of steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate based on disease imaging | From date of randomization until the date of first documented progression, assessed up to 63 weeks.
  Determine the objective response of GR-MD-02 + pembrolizumab versus pembrolizumab monotherapy in patients with advanced MM or HNSCC

SECONDARY OUTCOMES:
Evaluation of GAL-3 expression | Screening and Day 68
  Compare GAL-3 expression in paired biopsies after GR-MD-02 + pembrolizumab or pembrolizumab monotherapy.
Evaluation of predictive biomarker | Day 85
  Characterize MDSC expression over time as a predictive biomarker of response after GRMD02 + pembrolizumab or pembrolizumab monotherapy
Frequency of Immune-mediated adverse events | From time of informed consent to week 63
  Compare the frequency of immune-mediated adverse events after GR-MD-02 + pembrolizumab versus pembrolizumab + placebo
Evaluation of antiviral immunity | Day 85
  Assess the biological activity of GR-MD-02 + pembrolizumab and in comparison to pembrolizumab monotherapy by measuring CD4+T cells with a memory phenotype (CD3+CD4+Ki67+CD25+FoxP3-CCR7-CD45RA-CD27+CD28+/-).
Evaluation of antiviral immunity | Day 85
  Assess the biological activity of GR-MD-02 + pembrolizumab and in comparison to pembrolizumab monotherapy by measuring CD8+ T cells with effector phenotype (CD3+CD8+CD28-CD95+).
Evaluation of antiviral immunity | Day 85
  Assess the biological activity of GR-MD-02 + pembrolizumab and in comparison to pembrolizumab monotherapy by measuring tumor-specific T cells using autologous and/or HLA-matched tumor when available.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan D. Curti, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Portland Providence Medical Center, Portland, Oregon, United States